CLINICAL TRIAL: NCT02217098
Title: The Survival Rate of Glass Ionomer Cement, Glass Carbomer Cement and Compomer in Occlusal and Proximal ART Restorations
Acronym: ARTUSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Prócida Raggio (Other)
Collaborators: Academic Centre for Dentistry in Amsterdam (Other)
Responsible Party: Sponsor-Investigator, Daniela Prócida Raggio, Associated Professor of Paediatric Dentistry, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FOUSP6808912
Record Dates: First submitted 2014-05-21; First posted 2014-08-15 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Caries Involving Multiple Surfaces of Tooth; Dental Caries on Chewing Surface of Tooth; Dental Caries Extending Into Dentine
Keywords: ART; Occlusal; Occlusoproximal; Primary teeth
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GIC Restorations (Active Comparator): Restorations using Glass Ionomer Cement
  Interventions: Procedure: GIC Restorations
- Compomer Restorations (Experimental): Restorations using Compomer
  Interventions: Procedure: Compomer Restorations
- Carbomer Restorations (Experimental): Restorations using Glass Carbomer
  Interventions: Procedure: Carbomer Restorations

INTERVENTIONS:
Procedure: GIC Restorations — Restorations using Glass Ionomer Cement
  Arms: GIC Restorations
Procedure: Carbomer Restorations — Restorations using Glass Carbomer
  Arms: Carbomer Restorations
Procedure: Compomer Restorations — Restorations using Compomer
  Arms: Compomer Restorations

SUMMARY:
The null hypothesis of this study is that GCC, GIC and compomer have the same survival rate when used for the treatment of occlusal and proximal caries in primary molars with ART under field conditions.

This research will be done under field conditions in Barueri, a city in the state of São Paulo, Brazil. A total of 600 patients will be selected. After 1, 6, 12, 18 and 24 months the restorations and teeth will be evaluated by two independent evaluators. Only children whose parent or representative who have signed an informed consent are included in this research.The ART treatments will be done by two dental students. The operators will receive the same ART-training. The children will be randomly assigned to one of the operators. The restorative material to be used in each child will be assigned by another random list. It will be performed descriptive analyses to describe the sample. Bivariate analyses will be performed to test the hypothesis. The data will be analyzed with a chi-square test to compare the survival rates of GIC and GCC. Some co-variables will be evaluated, such as: operator effect, the influence of the cavity size on the survival rate, the position of the tooth, the dentists preferred side, the child's dmft/DMFT, contamination and finally the preoperative conditions. The effect of these variables on the survival rate will be evaluated using a regression analysis.

DETAILED DESCRIPTION:
The null hypothesis of this study is that GCC, GIC and compomer have the same survival rate when used for the treatment of occlusal and proximal caries in primary molars with ART under field conditions.

This research will be done under field conditions in Barueri, a city in the state of São Paulo, Brazil. A total of 600 patients will be selected, 300 patients with one occlusal carie lesion and 300 different patients with occlusal proximal cavities. After 1, 6, 12, 18 and 24 months the restorations and teeth will be evaluated by two independent evaluators. Only children whose parent or representative who have signed an informed consent are included in this research. Only one restoration per child will be included in this study. If more carious lesions are present, one of them will be randomly selected for this research. The remaining carious lesions will be also be treated. The ART treatments will be done by two dental students. The operators will receive the same ART-training.

The children will be randomly assigned to one of the operators. The restorative material to be used in each child will be assigned by another random list.

The selected children can have or an occlusal (O) cavity or an occlusalproximal (OP) cavity. So, the stratum of the study is OP and O. So, one randomization list will be performed for occlusal cavities and another randomization list will be used for occlusal proximal cavities.

It will be performed descriptive analyses to describe the sample. Bivariate analyses will be performed to test the hypothesis. The data will be analyzed with a chi-square test to compare the survival rates of GIC and GCC. Some co-variables will be evaluated, such as: operator effect, the influence of the cavity size on the survival rate, the position of the tooth, the dentists preferred side, the child's dmft/DMFT, contamination and finally the preoperative conditions. The effect of these variables on the survival rate will be evaluated using a regression analysis.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the patient:

* Healthy children, age: 4-8 years
* At least one occlusal or proximal carious lesion in primary molar involving dentin
* Cooperative behavior
* Presence of antagonist of the tooth

Inclusion criteria for the tooth:

* Carious lesion involving dentin with dimensions bucco-lingual and mesio-distal not greater than 2.5mm, occluso-cervical not greater than 2.0mm
* Absence of tooth mobility and abscess or fistula near to the selected tooth

Exclusion Criteria:

* Only children whose parent or representative who have signed an informed consent are included in this research. Only one restoration per child will be included in this study. If more carious lesions are present, one of them will be randomly selected for this research.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 530 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Survival rate (longevity) of ART restorations using differents materials | 6, 12, 24 and 36 months follow-up
  The null hypothesis of this study is that GCC, GIC and compomer have the same survival rate when used for the treatment of occlusal and occlusoproximal caries in primary molars with ART under field conditions.

SECONDARY OUTCOMES:
Association between survival and gender | 6, 12, 24 and 36 months follow-up
Association between survival and DMFT (caries experience) | 6, 12, 24 and 36 months follow-up
Association between survival and occlusal contact after restoration | 6, 12, 24 and 36 months follow-up
Association between sucess and ICDAS of the adjacent tooth (if there is a dentin cavited lesion or not) | 6, 12, 24 and 36 months follow-up
Cost-effectiveness of the 3 materials and their association with survival rate | 6, 12, 24 and 36 months follow-up
Comparition between Success of the restoration and longevity of the teeth (with or without pulp damage and exfoliation in the normal time) | 6, 12, 24 and 36 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Daniela P Raggio, Professor, Principal Investigator — Universidade de Sao Paulo - Faculdade de Odontologia; Isabel O Costa, PhD, Study Director — University of Sao Paulo
Locations (1):
- School of Dentistry - Sao Paulo University, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonifacio CC, Hesse D, Raggio DP, Bonecker M, van Loveren C, van Amerongen WE. The effect of GIC-brand on the survival rate of proximal-ART restorations. Int J Paediatr Dent. 2013 Jul;23(4):251-8. doi: 10.1111/j.1365-263X.2012.01259.x. Epub 2012 Aug 14. PMID 22891625
- [Background] de Amorim RG, Leal SC, Frencken JE. Survival of atraumatic restorative treatment (ART) sealants and restorations: a meta-analysis. Clin Oral Investig. 2012 Apr;16(2):429-41. doi: 10.1007/s00784-011-0513-3. Epub 2011 Jan 28. PMID 21274581
- [Background] Banerjee A, Kidd EA, Watson TF. In vitro evaluation of five alternative methods of carious dentine excavation. Caries Res. 2000 Mar-Apr;34(2):144-50. doi: 10.1159/000016582. PMID 10773632
- [Background] van Bochove JA, van Amerongen WE. The influence of restorative treatment approaches and the use of local analgesia, on the children's discomfort. Eur Arch Paediatr Dent. 2006 Mar;7(1):11-6. doi: 10.1007/BF03320809. PMID 17140522
- [Background] Carvalho TS, van Amerongen WE, de Gee A, Bonecker M, Sampaio FC. Shear bond strengths of three glass ionomer cements to enamel and dentine. Med Oral Patol Oral Cir Bucal. 2011 May 1;16(3):e406-10. doi: 10.4317/medoral.16.e406. PMID 20526266
- [Background] Cehreli SB, Tirali RE, Yalcinkaya Z, Cehreli ZC. Microleakage of newly developed glass carbomer cement in primary teeth. Eur J Dent. 2013 Jan;7(1):15-21. PMID 23408469
- [Background] Chen X, Du M, Fan M, Mulder J, Huysmans MC, Frencken JE. Effectiveness of two new types of sealants: retention after 2 years. Clin Oral Investig. 2012 Oct;16(5):1443-50. doi: 10.1007/s00784-011-0633-9. Epub 2011 Nov 29. PMID 22124610
- [Background] van Duinen RN, Kleverlaan CJ, de Gee AJ, Werner A, Feilzer AJ. Early and long-term wear of 'fast-set' conventional glass-ionomer cements. Dent Mater. 2005 Aug;21(8):716-20. doi: 10.1016/j.dental.2004.09.007. PMID 16026667
- [Background] Ersin NK, Candan U, Aykut A, Oncag O, Eronat C, Kose T. A clinical evaluation of resin-based composite and glass ionomer cement restorations placed in primary teeth using the ART approach: results at 24 months. J Am Dent Assoc. 2006 Nov;137(11):1529-36. doi: 10.14219/jada.archive.2006.0087. PMID 17082278
- [Background] Frencken JE, Pilot T, Songpaisan Y, Phantumvanit P. Atraumatic restorative treatment (ART): rationale, technique, and development. J Public Health Dent. 1996;56(3 Spec No):135-40; discussion 161-3. doi: 10.1111/j.1752-7325.1996.tb02423.x. PMID 8915958
- [Background] Kuhnisch J, Mansmann U, Heinrich-Weltzien R, Hickel R. Longevity of materials for pit and fissure sealing--results from a meta-analysis. Dent Mater. 2012 Mar;28(3):298-303. doi: 10.1016/j.dental.2011.11.002. Epub 2011 Dec 3. PMID 22137936
- [Background] Mickenautsch S, Mount G, Yengopal V. Therapeutic effect of glass-ionomers: an overview of evidence. Aust Dent J. 2011 Mar;56(1):10-5; quiz 103. doi: 10.1111/j.1834-7819.2010.01304.x. PMID 21332735
- [Background] Raggio DP, Hesse D, Lenzi TL, Guglielmi CA, Braga MM. Is Atraumatic restorative treatment an option for restoring occlusoproximal caries lesions in primary teeth? A systematic review and meta-analysis. Int J Paediatr Dent. 2013 Nov;23(6):435-43. doi: 10.1111/ipd.12013. Epub 2012 Nov 28. PMID 23190278
- [Derived] Olegario IC, Hesse D, Mendes FM, Bonifacio CC, Raggio DP. Glass carbomer and compomer for ART restorations: 3-year results of a randomized clinical trial. Clin Oral Investig. 2019 Apr;23(4):1761-1770. doi: 10.1007/s00784-018-2593-9. Epub 2018 Aug 31. PMID 30171345